CLINICAL TRIAL: NCT01191736
Title: Comparison of the Effectiveness of Ultra-Brief and Brief Hands-Only CPR Video Training With and Without Psychomotor Skill Practice for Lay Responders: a Controlled Randomized Study
Brief Title: Ultra-Brief Versus Brief Hands Only CPR Video Training With and Without Psychomotor Skill Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valleywise Health (Other)
Collaborators: American Heart Association (Other); University of Arizona (Other)
Responsible Party: Bentley J Bobrow, MD, FACEP, FAAEM, Maricopa Integrated Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009-070
Record Dates: First submitted 2010-08-27; First posted 2010-08-31 (Estimated); Results first posted 2010-10-07 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Cardiac Arrest
Keywords: hands only; CPR; resuscitation; cardiac arrest; Education of general public regarding resuscitation methods
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- No training, assessed within 60 mins (Experimental): Subjects receive no training
  Interventions: Behavioral: No training, assessed within 60 mins
- Ultra-brief video; assessed in 60 mins (Experimental): Subjects receive an ultra-brief (90-second) video on hands-only CPR
  Interventions: Behavioral: Ultra-brief video; assessed in 60 mins
- Brief video; assessed in 60 mins (Experimental): Subjects receive a brief (5-minute) video on hands-only CPR
  Interventions: Behavioral: Brief video; assessed in 60 mins
- Brief video + hands-on; ass'd in 60 mins (Experimental): Subjects receive a brief (5-minute) video with hands-on manikin practice
  Interventions: Behavioral: Brief video + hands-on; ass'd in 60 mins
- Ultra-brief video; assessed at 2 months (Experimental)
  Interventions: Behavioral: Ultra-brief video; assessed at 2 months
- Brief video; assessed 2 months later (Experimental)
  Interventions: Behavioral: Brief video; assessed 2 months later
- Brief video + hands-on; ass'd 2 ms later (Experimental)
  Interventions: Behavioral: Brief video + hands-on; ass'd 2 ms later

INTERVENTIONS:
Behavioral: No training, assessed within 60 mins — Subjects receive no training in resuscitation
  Other Names: C-Group
  Arms: No training, assessed within 60 mins
Behavioral: Ultra-brief video; assessed in 60 mins — Subjects receive an ultra-brief (90-second) video on hands-only CPR
  Other Names: UBV-Group
  Arms: Ultra-brief video; assessed in 60 mins
Behavioral: Brief video; assessed in 60 mins — Subjects receive a brief (5-minute) video on hands-only CPR
  Other Names: BV-Group
  Arms: Brief video; assessed in 60 mins
Behavioral: Brief video + hands-on; ass'd in 60 mins — Subjects receive a brief (5-minute) video with hands-on manikin practice
  Other Names: BVP-Group
  Arms: Brief video + hands-on; ass'd in 60 mins
Behavioral: Ultra-brief video; assessed at 2 months — Subjects see ultra-brief video (90-seconds), are assessed two months later
  Other Names: UBV-Group
  Arms: Ultra-brief video; assessed at 2 months
Behavioral: Brief video; assessed 2 months later — Subjects see brief video (5 minutes), are then assessed two months later
  Other Names: BV-Group
  Arms: Brief video; assessed 2 months later
Behavioral: Brief video + hands-on; ass'd 2 ms later — Subjects see brief (5-minute) video, receive hands-on training, and are assessed two months later
  Other Names: BVP-Group
  Arms: Brief video + hands-on; ass'd 2 ms later

SUMMARY:
Bystander CPR improves survival from Out of Hospital Cardiac Arrest. This study examines the efficacy of ultra-brief video training for Hands-Only CPR. Subjects were randomized to one of four training conditions, then assessed for CPR skills retention.

DETAILED DESCRIPTION:
Bystander CPR improves survival from Out of Hospital Cardiac Arrest. This study is the first of its kind to examine the efficacy of ultra-brief video training for Hands-Only CPR without the use of a manikin. The results will inform future efforts to mass train citizens in CPR. Subjects were randomized to one of four training conditions, then assessed for CPR skills retention. The four groups were 1) no training; 2) ultra-brief training video (90 seconds); 3) short training video (5 minutes) with no practice; and 4) short training video with hands-on practice. The subjects were then evaluated for CPR skills retention. One half of the subjects were evaluated on the training day, and the other half were evaluated two months later.

ELIGIBILITY:
Inclusion Criteria:

* Members of a local area church

Exclusion Criteria:

* Less than 18 years old
* formal CPR training or certification within last 2 years
* Lacks fluency in English
* Works as a health care provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bentley J Bobrow, MD, Principal Investigator — Valleywise Health

REFERENCES:
- [Derived] Bobrow BJ, Vadeboncoeur TF, Spaite DW, Potts J, Denninghoff K, Chikani V, Brazil PR, Ramsey B, Abella BS. The effectiveness of ultrabrief and brief educational videos for training lay responders in hands-only cardiopulmonary resuscitation: implications for the future of citizen cardiopulmonary resuscitation training. Circ Cardiovasc Qual Outcomes. 2011 Mar;4(2):220-6. doi: 10.1161/CIRCOUTCOMES.110.959353. Epub 2011 Mar 8. PMID 21386066

RESULTS

PARTICIPANT FLOW:
Groups:
- No Training, Assessed Within 60 Mins: The subjects received no training and were assessed within 60 minutes
- Ultra-brief Video; Assessed at 2 Months: Subjects receive an ultra-brief (90-second) video on hands-only CPR, and were assessed 2 months later
- Brief Video; Assessed 2 Months Later: Subjects receive a brief (5-minute) video on hands-only CPR, and were assessed two months later
- Brief Video + hands-on; Ass'd 2 Months Later: Subjects receive a brief (5-minute) video with hands-on manikin practice, and were assessed 2 months later
Period: Overall Study
Arm/Group | No Training, Assessed Within 60 Mins | Ultra-brief Video; Assessed in 60 Mins | Brief Video; Assessed in 60 Mins | Brief Video + hands-on; Ass'd in 60 Mins | Ultra-brief Video; Assessed at 2 Months | Brief Video; Assessed 2 Months Later | Brief Video + hands-on; Ass'd 2 Months Later
Started | 51 | 47 | 49 | 46 | 48 | 50 | 45
Completed | 51 | 47 | 49 | 46 | 48 | 50 | 45
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Training, Assessed Within 60 Mins | Ultra-brief Video; Assessed in 60 Mins | Brief Video; Assessed in 60 Mins | Brief Video + hands-on; Ass'd in 60 Mins | Ultra-brief Video; Assessed at 2 Months | Brief Video; Assessed 2 Months Later | Brief Video + hands-on; Ass'd 2 Months Later | Total
Number analyzed (Participants) | 51 | 47 | 49 | 46 | 48 | 50 | 45 | 336
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 0 | 3 | 0 | 2 | 0 | 7
  Between 18 and 65 years | 48 | 32 | 41 | 39 | 43 | 44 | 42 | 289
  >=65 years | 2 | 14 | 8 | 4 | 5 | 4 | 3 | 40
Age Continuous [Mean (Standard Deviation); unit: years] | 44.8 (11.8) | 51.7 (15.2) | 50.5 (13.3) | 41.7 (14.2) | 48.1 (14.5) | 45.3 (13.8) | 47.4 (11.9) | 47.1 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 22 | 29 | 22 | 27 | 25 | 181
  Male | 23 | 19 | 27 | 17 | 26 | 23 | 20 | 155
Region of Enrollment [Number; unit: participants]
  United States | 51 | 47 | 49 | 46 | 48 | 50 | 45 | 336

OUTCOME MEASURES:

1. Primary Outcome: Median Compression Depth (mm)
Description: Assessment of resuscitation skills using a Laerdal Resusci Annie recording manikin and Laerdal PC Skill Reporting software
Time Frame: 60 minutes after intervention or two months after intervention
Population: Per protocol
Measure: Median (Inter-Quartile Range); unit: millimeters
Arm/Group | No Training, Assessed Within 60 Mins | Ultra-brief Video; Assessed in 60 Mins | Brief Video; Assessed in 60 Mins | Brief Video + hands-on; Ass'd in 60 Mins | Ultra-brief Video; Assessed at 2 Months | Brief Video; Assessed 2 Months Later | Brief Video + hands-on; Ass'd 2 Months Later
Number analyzed (Participants) | 51 | 47 | 49 | 46 | 48 | 50 | 45
millimeters | 30 [14 to 41] | 41 [32 to 51] | 42 [34 to 51] | 48 [39 to 55] | 43 [30 to 49] | 43 [32 to 55] | 46 [32 to 55]
Statistical Analysis 1: Comparison: No Training, Assessed Within 60 Mins vs Ultra-brief Video; Assessed in 60 Mins vs Brief Video; Assessed in 60 Mins vs Brief Video + hands-on; Ass'd in 60 Mins vs Ultra-brief Video; Assessed at 2 Months vs Brief Video; Assessed 2 Months Later vs Brief Video + hands-on; Ass'd 2 Months Later; Kruskal-Wallis test for multiple comparisons; Test type: Superiority or Other; p = .05, Kruskal-Wallis; Null hypothesis: the medians for all seven arms are equal

2. Secondary Outcome: The Proportion of Subjects Who Assessed the Responsiveness of the Victim (Manikin) as Judged by Expert Raters
Description: The proportion of the subjects who assessed the responsiveness of the victim (manikin) as judged by expert raters
Time Frame: 60 minutes after intervention and two months after intervention
Measure: Mean (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | No Training, Assessed Within 60 Mins | Ultra-brief Video; Assessed in 60 Mins | Brief Video; Assessed in 60 Mins | Brief Video + hands-on; Ass'd in 60 Mins | Ultra-brief Video; Assessed at 2 Months | Brief Video; Assessed 2 Months Later | Brief Video + hands-on; Ass'd 2 Months Later
Number analyzed (Participants) | 51 | 47 | 49 | 46 | 48 | 50 | 45
Proportion of Participants | .854 [.754 to .954] | .182 [.068 to .296] | .8 [.683 to .917] | .978 [.936 to 1.000] | .542 [.401 to .683] | .780 [.665 to .895] | .822 [.711 to .934]
Statistical Analysis 1: Comparison: No Training, Assessed Within 60 Mins vs Ultra-brief Video; Assessed in 60 Mins vs Brief Video; Assessed in 60 Mins vs Brief Video + hands-on; Ass'd in 60 Mins vs Ultra-brief Video; Assessed at 2 Months vs Brief Video; Assessed 2 Months Later vs Brief Video + hands-on; Ass'd 2 Months Later; Comparison of proportions of subjects who assessed responsiveness; Test type: Superiority or Other; p = .05, Chi-squared; Null hypothesis: the proportions within the seven arms are equal

ADVERSE EVENTS:
Description: In this study, the subjects practice CPR methods on a manikin. There really is no risk to the subjects. Therefore the number of subjects exposed to a risk is zero for each of the seven arms, and zero overall.
Arm/Group | No Training, Assessed Within 60 Mins | Ultra-brief Video; Assessed in 60 Mins | Brief Video; Assessed in 60 Mins | Brief Video + hands-on; Ass'd in 60 Mins | Ultra-brief Video; Assessed at 2 Months | Brief Video; Assessed 2 Months Later | Brief Video + hands-on; Ass'd 2 Months Later
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes